CLINICAL TRIAL: NCT06377228
Title: A Phase 1b, Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of TAK-007, an Allogeneic Anti-CD19 Chimeric Antigen Receptor Natural Killer Cell (CD19 CAR-NK) Therapy, in Adult Subjects With Refractory Lupus Nephritis or Refractory Systemic Sclerosis
Brief Title: A Study of TAK-007 in Adults With Refractory Lupus Nephritis (LN) or Refractory Systemic Sclerosis (SSc)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision (no safety concerns)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-007-1001
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Refractory Lupus Nephritis; Refractory Systemic Sclerosis
Keywords: Drug Therapy
MeSH Terms: conditions — Lupus Nephritis; Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LN Cohort: Single Dose TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells (Experimental): Participants with LN will receive IV LDC, for 3 days in conditioning phase (Days -5, -4, and -3), followed by a single dose of IV 800 × 10^6 TAK-007 on Day 1 with a potential to explore an alternate dose level if deemed appropriate.
  Interventions: Biological: TAK-007; Drug: Chemotherapy Agents
- SSc Cohort: Part 1a: Single Dose TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells (Experimental): Participants with SSc will receive IV LDC, for 3 days in conditioning phase (Days -5, -4, and -3), followed by a single dose of IV 800 × 10^6 TAK-007 on Day 1.
  Interventions: Biological: TAK-007; Drug: Chemotherapy Agents
- SSc Cohort: Part 1b: Multiple Dose TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells (Experimental): Participants with SSc will receive IV LDC, for 3 days in conditioning phase (Days -5, -4, and -3), followed by multiple doses of IV 800 × 10^6 TAK-007 on Days 1, 8, and 15.
  Interventions: Biological: TAK-007; Drug: Chemotherapy Agents
- SSc Cohort: Part 2 (Dose Expansion): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells (Experimental): Based on the data of Part 1, Part 2 may be initiated for participants with SSc to receive IV LDC, for 3 days in conditioning phase (Days -5, -4, and -3), followed by either single dose of IV 800 × 10^6 TAK-007 on Day 1 or multiple doses of IV 800 × 10^6 TAK-007 on Days 1, 8, and 15.
  Interventions: Biological: TAK-007; Drug: Chemotherapy Agents

INTERVENTIONS:
Biological: TAK-007 — TAK-007 IV infusion.
Drug: Chemotherapy Agents — Fludarabine and cyclophosphamide IV infusion.

SUMMARY:
The main aim of the trial is to learn how well adults with refractory lupus nephritis (LN) or refractory systemic sclerosis (SSc) tolerate TAK-007 and to check for side effects (adverse events).

Other aims are to learn how effective treatment with TAK-007 is in adults with refractory LN or refractory SSc, what effects TAK-007 has on the human body, and whether participants will produce antibodies against TAK-007.

DETAILED DESCRIPTION:
The drug being tested in this trial is called TAK-007. TAK-007 is being tested to treat people with refractory LN or refractory SSc. This trial will look at the safety and tolerability of TAK-007.

The trial will enroll approximately 26 participants. Participants will receive a single dose or multiple doses of TAK-007, which is an anti-CD19 chimeric antigen receptor natural killer cell (CD19 CAR-NK) therapy.

Participants with refractory LN will be treated with 3 days of intravenous (IV) lymphodepleting chemotherapy (LDC) and then after a gap of at least 2 days, a single IV dose of TAK-007 on Day 1. For participants with refractory SSc the trial has 2 parts. In Part 1, participants with refractory SSc will be treated with 3 days of IV LDC and then after a gap of at least 2 days, a single IV dose (Part 1a - single dose) or three IV doses (Part 1b - multiple doses) of TAK-007. Based on the data of Part 1, Part 2 (expansion) may be initiated in participants with refractory SSc to further evaluate the impact of LDC followed by single dose or multiple doses of TAK-007.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is approximately 24 months.

ELIGIBILITY:
Inclusion Criteria for LN Cohort:

1. The participant must have a diagnosis of SLE fulfilling European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) 2019 classification criteria.
2. The participant must have a histologically proven glomerulonephritis (proliferative LN class III or IV, with or without the presence of class V, according to 2018 International Society of Nephrology/Renal Pathology Society [ISN/RPS] criteria).
3. The participant must be positive for ANA at screening or by documented medical history, and at least one of the following autoantibodies at screening: anti-dsDNA or anti-Smith (Sm) antibody.
4. The participant has had an inadequate response, defined as failure to improve within 12 weeks, based on investigator discretion, to at least 2 standard-of-care treatments for SLE (including glucocorticoids and immunosuppressive agents) OR at least 1 biologic treatment for SLE.
5. The participant has a SLEDAI-2K total score ≥6.

   Inclusion Criteria for SSc Cohort:
6. The participant must have a diagnosis of SSc fulfilling EULAR/ACR 2013 classification criteria.
7. The participant must have an early disease: 5 years or less of disease duration since first non-Raynaud's sign or symptom.
8. The participant must have evidence for presence of Interstitial Lung Disease (ILD) on HRCT imaging.
9. The participant must have active disease.
10. Positive for ANA (by immunofluorescent assay [IFA] with a titer ≥1:80) at screening or by documented medical history.
11. Lack of response or insufficient response (based on investigator discretion), to adequate doses of at least one of the following treatments used for at least 4 months: cyclophosphamide, methotrexate, mycophenolate (MMF)/mycophenolic acid, nintedanib, rituximab, or tocilizumab. Intolerance is not considered an insufficient response.

    Inclusion Criteria for LN and SSc Cohorts:
12. The participant must have adequate bone marrow function.
13. The participant must have adequate renal, hepatic, cardiac, and pulmonary function.
14. The participant is willing and able to understand and fully comply with trial procedures and requirements in the opinion of the investigator.
15. The participant has provided informed consent and any required privacy authorization before the initiation of any trial procedures.
16. The participant must be aged 18 to 75 years (inclusive) at the time of consent.
17. Participants with female reproductive anatomy must be:

    1. postmenopausal for at least 1 year before the screening visit, OR
    2. surgically sterile for at least 6 weeks, OR
    3. if the participant is of childbearing potential, must:

    i. Agree to practice 1 highly effective method of contraception and 1 additional effective (barrier) method at the same time, from the time of signing the informed consent through at least 24 months following TAK-007 administration OR ii. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant (periodic abstinence [for example, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception). Female and male condoms should not be used together AND iii. Agree not to donate an egg or eggs (ova) or breastfeed a baby during the trial and until at least 24 months following TAK-007 administration.
18. Participants with male reproductive anatomy, even if surgically sterilized (that is, status post vasectomy), must:

    1. Agree to practice effective barrier contraception from the time of signing the informed consent through at least 6 months following TAK-007 administration, or
    2. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant (periodic abstinence [for example, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception), and
    3. Agree not to donate sperm during the trial and at least 6 months following TAK-007 administration.

Exclusion Criteria for LN Cohort:

1. The participant has a history of drug-induced SLE.
2. The participant has a current diagnosis of active or unstable neuropsychiatric lupus (e.g., cerebritis, cerebrovascular accident, and seizures). However, participants with mononeuritis multiplex or polyneuropathy can be included in the study.
3. The participant has a history of catastrophic antiphospholipid syndrome or saddle embolism (antiphospholipid syndrome adequately controlled by anticoagulant therapy for at least 3 months is acceptable).
4. The participant has a history or current diagnosis of other autoimmune diseases or current inflammatory joint or skin disease other than SLE that, in the opinion of the investigator and per sponsor assessment, could interfere with the inflammatory arthritis or skin assessments and confound the disease activity assessments.

   Exclusion Criteria for SSc Cohort:
5. The participant has ppFVC ≤45% or DLCO ≤40% or requiring supplemental oxygen at screening.
6. The participant has pulmonary arterial hypertension requiring active treatment.
7. The participant has anti-centromere antibody.
8. The participant has a history of severe scleroderma renal crisis OR scleroderma renal crisis within 6 months prior to Day 1.
9. The participant has obstructive pulmonary disease (pre-bronchodilator forced expiratory volume in 1 second (FEV1)/FVC <0.7)
10. The participant has significant emphysema on screening HRCT, based on qualitative investigator assessment (extent of emphysema exceeds extent of ILD).
11. The participant has a history or current diagnosis of other systemic autoimmune diseases or current inflammatory joint or skin disease other than SSc that, in the opinion of the investigator and per sponsor assessment, could interfere with the trial assessments and confound the disease activity assessments.
12. The participant has actively bleeding gastric antral vascular ectasia
13. The participant has severe SSc-related lower gastrointestinal involvement requiring nutrition via percutaneous endoscopic gastrostomy/percutaneous endoscopic jejunostomy (PEG/PEJ) tube or parental nutrition.

    Exclusion Criteria for Both LN and SSc Cohorts:
14. The participant has any clinically significant medical condition, evidence of an unstable clinical condition (for example, cardiovascular, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, or immunologic), or vital signs/physical/laboratory/electrocardiogram (ECG) abnormality that would, in the opinion of the investigator and per sponsor assessment, put the participant at undue risk or interfere with interpretation of trial results.
15. The participant has a history of active infection (for example, coronavirus disease 2019 [COVID-19], influenza) or febrile illness within 7 days before enrollment.
16. Viral diseases:

    1. The participant is positive for hepatitis C virus (HCV) antibody and has a positive confirmatory test result for HCV ribonucleic acid [RNA] (nucleic acid test or polymerase chain reaction [PCR]).
    2. The participant is positive for hepatitis B surface antigen, hepatitis B virus (HBV) deoxyribonucleic acid (DNA), or hepatitis B core antibody.
    3. The participant has a history of human immunodeficiency virus (HIV) infection or has positive serology for HIV.
17. The participant has a history of significant chronic or recurrent bacterial disease, including but not limited to chronic pyelonephritis or cystitis, chronic bronchitis/pneumonitis, osteomyelitis, chronic skin ulcerations/infections or fungal infections, or latent tuberculosis infection.
18. The participant has a known or suspected allergy to TAK-007, or any of its components, or to cyclophosphamide or fludarabine.
19. The participant is unable to comply with the restrictions and prohibited treatments and/or discontinuation requirements.
20. The participant has given greater than 500 mL of blood or plasma within 30 days of screening (during a clinical trial or at a blood bank donation) or plans to donate blood during the course of the trial.
21. The participant is compulsorily detained for treatment of either a psychiatric or physical (for example, infectious disease) illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-13 (Estimated); Primary Completion 2030-09-02 (Estimated); Study Completion 2030-09-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From first dose of LDC up to end of study (EOS) [up to Month 24]
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. TEAEs are defined as any AE that begins on or after the start date of LDC.
Number of Participants With Dose Limiting Toxicities (DLTs) | Up to Day 30
  DLTs are defined as any event throughout the study meeting the protocol-defined criteria that occur by Day 30 after administration of TAK-007 infusion on Day 1.

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for TAK-007 | Pre-dose and at multiple time points post-dose up to Month 24
Tmax: Time to Reach the Cmax for TAK-007 | Pre-dose and at multiple time points post-dose up to Month 24
Tlast: Time of Last Measurable Concentration Above the Lower Limit of Quantitation for TAK-007 | Pre-dose and at multiple time points post-dose up to Month 24
AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-007 | Pre-dose and at multiple time points post-dose up to Month 24
Change From Baseline in CD19+ B Cell Counts | Baseline up to Month 24
Change From Baseline in Plasma Cytokine Levels | Baseline up to Month 3
Change From Baseline in Clinician's Global Assessment (CGA) Score | Baseline up to Month 24
  The CGA score is a visual analogue score that reflects a clinician's judgement of overall systemic lupus erythematosus (SLE) activity. The CGA score ranges from 0 (none) to 3 (severe). Higher score indicates more severe disease activity.
Percentage of Participants With Antidrug Antibodies Categorized as Anti-Human Leukocyte Antigen (HLA) and Anti- Chimeric Antigen Receptor (CAR) | Up to Month 24
Percentage of Participants With Replication Competent Retrovirus (RCR) in Blood | Up to Month 24
Percentage of Participants With Refractory LN Achieving a Reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) Relative to Baseline | Baseline through Month 24
  The SLEDAI-2K is a measure of global disease activity in systemic lupus erythematosus. It consists of 24 weighted clinical and laboratory variables. The scores of the descriptors range from 1 to 8, and the total possible score for all 24 descriptors is 105, with higher scores representing increased disease activity.
Percentage of Participants With Refractory LN Achieving Complete Renal Response (CRR) | Up to Month 24
  CRR is defined as the fulfilment of following criteria: Ratio of urinary protein to creatinine of less than (<)0.5 mg/mg; ; Estimated glomerular filtration rate (eGFR) that was no worse than 10 percent (%) below the pre-flare value or greater than or equal to (≥)60 milliliters (mL) per minute per 1.73 meter^2 (m^2); No use of rescue therapy.
Time to CRR in Participants With Refractory LN | Up to Month 24
  CRR is defined as the fulfilment of following criteria: ratio of urinary protein to creatinine of <0.5 mg/mg; eGFR that was no worse than 10% below the pre-flare value or ≥60 mL per minute per 1.73 m^2; No use of rescue therapy.
Duration of CRR in Participants With Refractory LN | Up to Month 24
  CRR is defined as the fulfilment of following criteria: ratio of urinary protein to creatinine of <0.5 mg/mg; eGFR that was no worse than 10 % below the pre-flare value or ≥60 mL per minute per 1.73 m^2; No use of rescue therapy.
Percentage of Participants With Refractory LN Achieving Lupus Low Disease Activity State (LLDAS) | Up to Month 24
  The LLDAS is defined as: SLEDAI-2K less than or equal to (≤)4, with no activity in major organ systems (renal, central nervous system (CNS), cardiopulmonary, vasculitis, fever) and no hemolytic anemia or gastrointestinal activity; no new lupus disease activity compared with the previous assessment; a Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA)-SLEDAI physician global assessment (scale 0-3) ≤1; a current prednisolone (or equivalent) dose ≤7.5 milligrams (mg) daily; and well-tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents.
Time to LLDAS in Participants With Refractory LN | Up to Month 24
  The LLDAS is defined as: SLEDAI-2K ≤4, with no activity in major organ systems (renal, CNS, cardiopulmonary, vasculitis, fever) and no hemolytic anemia or gastrointestinal activity; no new lupus disease activity compared with the previous assessment; a SELENA-SLEDAI physician global assessment (scale 0-3) ≤1; a current prednisolone (or equivalent) dose ≤7.5 mg daily; and well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents.
Duration of LLDAS in Participants With Refractory LN | Up to Month 24
  The LLDAS is defined as: SLEDAI-2K ≤4, with no activity in major organ systems (renal, CNS, cardiopulmonary, vasculitis, fever) and no hemolytic anemia or gastrointestinal activity; no new lupus disease activity compared with the previous assessment; a SELENA-SLEDAI physician global assessment (scale 0-3) ≤1; a current prednisolone (or equivalent) dose ≤7.5 mg daily; and well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents.
Percentage of Participants With Refractory LN Meeting the Definition of Remission in Systemic Lupus Erythematosus (DORIS) Criteria | Up to Month 24
  DORIS remission is defined as achieving a SLEDAI-2K = 0 and a physician's global assessment score (PGA) <0.5, irrespective of serology, with permitted use of antimalarials, low-dose glucocorticoids (prednisolone ≤5 mg/day), and/or stable immunosuppressives and biologics.
Time to DORIS Remission in Participants With Refractory LN | Up to Month 24
  DORIS remission is defined as achieving a SLEDAI-2K = 0 and a PGA <0.5, irrespective of serology, with permitted use of antimalarials, low-dose glucocorticoids (prednisolone ≤5 mg/day), and/or stable immunosuppressives and biologics.
Duration of DORIS Remission in Participants With Refractory LN | Up to Month 24
  DORIS remission is defined as achieving a SLEDAI-2K = 0 and a PGA <0.5, irrespective of serology, with permitted use of antimalarials, low-dose glucocorticoids (prednisolone ≤5 mg/day), and/or stable immunosuppressives and biologics.
Change From Baseline in Anti-Double Stranded Deoxyribonucleic Acid (Anti-dsDNA) Levels in Participants With Refractory LN | Baseline up to Month 24
Change From Baseline in Antinuclear Antibody (ANA) Levels in Participants With Refractory LN | Baseline up to Month 24
Change From Baseline in Proteinuria Levels in Participants With Refractory LN | Baseline up to Month 24
Change From Baseline in Serum Creatinine Levels in Participants With Refractory LN | Baseline up to Month 24
Change From Baseline in eGFR in Participants With Refractory LN | Baseline up to Month 24
Change From Baseline in Complement (C3, C4) Levels in Participants With Refractory LN | Baseline up to Month 24
Change From Baseline in Forced Vital Capacity (FVC) in Participants With Refractory SSc | Baseline up to Month 24
  FVC (measured in mL) is defined as the maximal volume of air exhaled with maximally forced expiratory effort from a position of maximal inspiration.
Change From Baseline in Percentage (%) Predicted Forced Vital Capacity (ppFVC) in Participants With Refractory SSc | Baseline up to Month 24
Percentage of Refractory SSc Participants With no Worsening of Pulmonary Function | Up to Month 24
  Worsening of pulmonary function is defined as a decline from baseline in ppFVC greater than (>)3% predicted.
Change From Baseline in Adjusted Carbon Monoxide Diffusing Capacity (DLCO) % Predicted in Participants With Refractory SSc | Baseline up to Month 24
Change From Baseline in Modified Rodnan Skin Score (mRSS) in Participants With Refractory SSc | Baseline up to Month 24
  mRSS is a measure to assess skin thickness through skin palpation. The score is based on a scale of 0 to 3 which examines 17 body areas where 0 indicates no thickening of skin and 3 indicates severe thickening. Total mRSS ranges from 0 (best possible outcome) to 51 (worst possible outcome).
Change From Baseline in Patient Global Assessment (PtGA) in Participants With Refractory SSc | Baseline up to Month 24
  PtGA assesses participant's perception regarding the severity of their disease activity. The PtGA is a visual analog scale (VAS) measuring 100 millimeters (mm) in length. The participant marks on the line the value they feel best reflects their current overall SSc activity. The PtGA VAS is anchored with 0 on the left and 10 on the right, where 10 is maximal activity. Lower scores denote improvement.
Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) in Participants With Refractory SSc | Baseline up to Month 24
  HAQ-DI is a patient-reported questionnaire which consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants will assess their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task will be summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three=very severe, high-dependency disability.
Percentage of Participants Achieving Revised Composite Response Index in Systemic Sclerosis (R-CRISS) Response | Up to Month 24
  R-CRISS is used to categorize participants as responders or non-responders based on improvement or worsening in applicable components.
Change From Baseline in Quantitative Interstitial Lung Disease Score in the Whole Lung (QILD-WL) on High-Resolution Computed Tomography (HRCT) Scan of the Thorax in Participants With Refractory SSc | Baseline up to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/